CLINICAL TRIAL: NCT06638853
Title: The STRIDE Study (Strengthening Tolerance and Resilience in Dealing with Emotions): Pilot Testing of a School-Based Distress Tolerance Skills Program for Reducing Risk of Psychopathology in Adolescence
Brief Title: Piloting a School-Based Distress Tolerance Skills Program for Adolescents
Acronym: STRIDE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: Valley Catholic Middle School (Unknown)
Responsible Party: Principal Investigator, Bonnie Nagel, Principal Investigator, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00027611
Record Dates: First submitted 2024-10-09; First posted 2024-10-15 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2024-10

CONDITIONS: Distress, Emotional; Internalizing Mental Health Symptoms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Distress Tolerance Skills Training (Experimental): Students will participate in a series of classroom-based lessons aimed at increasing distress tolerance.
  Interventions: Behavioral: Distress Tolerance Skills Training
- Standard Curriculum (Control) (No Intervention): Students will not participate in the distress tolerance skills training. They will receive only their standard curriculum during class time.

INTERVENTIONS:
Behavioral: Distress Tolerance Skills Training — These lessons are adapted from "DBT Skills in Schools: Skills Training for Emotional Problem Solving for Adolescents (DBT STEPS-A)" by Mazza et al. and include elements of mindfulness training, psychoeducation about emotions, and techniques/skills for managing extreme emotions.
  Arms: Distress Tolerance Skills Training

SUMMARY:
Research suggests that an individual's perceived ability to withstand distressing or upsetting emotions (i.e., distress tolerance; DT) is a common risk factor across several mental health conditions that commonly emerge during adolescence. This study aims to evaluate the acceptability, feasibility, and initial efficacy of a classroom-based DT skills training program for middle school students. This study will also explore associations between changes in DT and internalizing symptoms (e.g., anxiety, depression).

DETAILED DESCRIPTION:
A variety of deleterious mental health conditions have their peak age of onset in adolescence, including depression and anxiety. Distress tolerance (DT) - defined as the perceived or actual ability to withstand aversive emotional states - has been postulated as a transdiagnostic risk factor across several "emotional" disorders that typically emerge during adolescence. Importantly, while there is compelling evidence that DT is associated with emotion dysregulation and symptom severity, it is unclear whether modifying DT can reduce future risk for psychopathology in adolescent populations. This proposal aims to evaluate the feasibility, acceptability, and initial efficacy of a classroom-based DT intervention for middle school students. Additionally, this proposal will examine associations between changes in DT and internalizing symptoms.

Primary Objective:

To evaluate the acceptability, feasibility, and efficacy of a classroom-based DT skills training program for middle school students.

Secondary Objectives:

To examine whether participation in the DT skills training program is associated with lower severity of internalizing symptoms over the course of the academic year.

ELIGIBILITY:
Inclusion Criteria:

* Middle school aged-youth attending Valley Catholic Middle School in grade 6, 7, or 8

Exclusion Criteria:

* None

Ages: 11 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 74 (Actual)
Dates: Start 2024-10-25 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Feasibility | Pre-intervention and immediately post-intervention
  Consent rates during enrollment and attrition rates during the study will be used to assess the feasibility of the intervention.
Acceptability | Immediately post-intervention
  The investigators will use a brief feedback survey at the end of the study to gather information about participants' experiences of the intervention. Responses on this survey will be used to determine the acceptability of the intervention.
Distress Tolerance | Pre-intervention, immediately post-intervention, 3-month follow-up, and 6-month follow-up
  The investigators will assess change in distress tolerance from pre-intervention to post-intervention. Distress tolerance will be indexed by total scores on the Distress Tolerance Scale (DTS), which is a 15-item self-report measure that assesses the respondent's perceived ability to withstand distressing or upsetting emotional states. Possible total scores can range from 15 to 75. Higher scores indicate higher distress tolerance. This outcome measure will be examined and compared for both the intervention group and the control group.

SECONDARY OUTCOMES:
Internalizing Symptoms | Pre-intervention, immediately post-intervention, 3-month follow-up, and 6-month follow-up
  The investigators will assess change in internalizing symptoms from pre-intervention to post-intervention and periodically during follow-up. Internalizing symptoms will be measured using the ASEBA Youth Self-Report (YSR). Possible raw scores on the Internalizing Symptoms Subscale can range from 0 to 62. Raw scores are transformed to standardized T-scores normed by age and gender and can range from 26 to 100. Higher scores indicate greater symptoms. This outcome measure will be examined and compared for both the intervention group and the control group.

CONTACTS AND LOCATIONS:
Overall Officials: Bonnie Nagel, PhD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Valley Catholic Middle School, Beaverton, Oregon, United States

IPD SHARING:
Plan to Share IPD: No